CLINICAL TRIAL: NCT05969171
Title: A Single-center, Prospective, Two Cohort Study of Surufatinib Combined With Gemcitabine and Nab-paclitaxel or Gemcitabine Combined With Nab-paclitaxel in the First-line Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Single-center, Prospective, Two Cohort Study of Surufatinib Combined With AG or AG in the First-line Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jin Xu, Director of Pancreatic Surgery, Fudan University ShangHai Cancer Center, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SH-PC101
Record Dates: First submitted 2023-06-08; First posted 2023-08-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Metastatic
MeSH Terms: interventions — surufatinib; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib in combination with gemcitabine and nab-paclitaxel (Experimental): Nab-paclitaxel: 125mg/m2 intravenously, d1, 8; every 3 weeks for a treatment cycle, did not exceed a maximum of 6 treatment cycles.
  Gemcitabine: 1000mg/m2, intravenous infusion greater than 30min, d1, 8, every 3 weeks for a treatment cycle.
  Surufatinib: 250mg, qd, po, every 3 weeks for a treatment cycle. Surufatinib and gemcitabine was continued until disease progression (PD, RECIST 1.1) or death (while the patient was on treatment) or toxicity became intolerant or other criteria for discontinuation of study therapy were met in the protocol. Allow adjustment of dosage according to protocol requirements, including suspension, lowering of dosage or permanent discontinuation.
  Interventions: Drug: Surufatinib, gemcitabine, nab-paclitaxel
- Nab-paclitaxel combined with gemcitabine (Active Comparator): Nab-paclitaxel: 125mg/m2 intravenously, d1, 8; every 3 weeks as a treatment cycle, should not exceed a maximum of 6 treatment cycles.
  Gemcitabine: 1000mg/m2, intravenous infusion greater than 30min, d1, 8, every 3 weeks as a treatment cycle, treatment until toxicity intolerance or disease progression, death, or other criteria for termination of study therapy as specified in the protocol.
  Allow adjustment of dosage according to protocol requirements, including suspension, lowering of dosage or permanent discontinuation.
  Interventions: Drug: Nab-paclitaxel, gemcitabine

INTERVENTIONS:
Drug: Surufatinib, gemcitabine, nab-paclitaxel — Nab-paclitaxel: 125mg/m2 intravenously, d1, 8; every 3 weeks for a treatment cycle, did not exceed a maximum of 6 treatment cycles. Gemcitabine: 1000mg/m2, intravenous infusion greater than 30min, d1, 8, every 3 weeks for a treatment cycle. Surufatinib: 250mg, qd, po, every 3 weeks for a treatment cycle. Surufatinib and gemcitabine was continued until disease progression (PD, RECIST 1.1) or death (while the patient was on treatment) or toxicity became intolerant or other criteria for discontinuation of study therapy were met in the protocol. Allow adjustment of dosage according to protocol requirements, including suspension, lowering of dosage or permanent discontinuation.
  Arms: Surufatinib in combination with gemcitabine and nab-paclitaxel
Drug: Nab-paclitaxel, gemcitabine — Nab-paclitaxel: 125mg/m2 intravenously, d1, 8; every 3 weeks as a treatment cycle, should not exceed a maximum of 6 treatment cycles. Gemcitabine: 1000mg/m2, intravenous infusion greater than 30min, d1, 8, every 3 weeks as a treatment cycle, treatment until toxicity intolerance or disease progression, death, or other criteria for termination of study therapy as specified in the protocol. Allow adjustment of dosage according to protocol requirements, including suspension, lowering of dosage or permanent discontinuation.
  Arms: Nab-paclitaxel combined with gemcitabine

SUMMARY:
This is a single-center, prospective, two cohort study to evaluate the efficacy and safety of surufatinib in combination with AG or AG alone in the first-line treatment of patients with locally advanced or metastatic pancreatic cancer.

Participants with previously received AG chemotherapy for 2 cycles with no disease progression will be enrolled:

Arm 1: Surufatinib plus AG chemotherapy (q3w) until disease progression/death/withdrawn; Arm 2: AG chemotherapy (q3w) until disease progression/death/withdrawn;

During the treatment period, imaging methods were used to evaluate the tumor status every 6 weeks (±7 days) until disease progression (RECIST 1.1) or death (during the patient's treatment) or toxicity was intolerable or other criteria for termination of study treatment specified in the protocol were met, and the tumor treatment and survival status after disease progression were recorded. Safety observation indicators include: AEs, changes in laboratory values, vital signs, and changes in electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria for enrollment:

1. The subjects voluntarily joined the study and signed the informed consent with good compliance and follow-up;
2. Unresectable, locally advanced or metastatic pancreatic cancer confirmed by histopathology or cytology;
3. Aged between 18 and 75 (including 18 and 75), male or female;
4. ECOG score: 0-1; Expected survival ≥12 weeks;
5. Patients who had previously received 2 cycles of AG regimen first-line systemic therapy for locally advanced or metastatic pancreatic cancer and whose efficacy was evaluated as CR, PR, SD (excluding SD patients whose efficacy was evaluated as increased after 2 cycles of therapy);
6. Patients with postoperative distant metastasis had received adjuvant chemotherapy of one type and the distance from adjuvant therapy time > Patients with recurrence at 6 months could be included in the group;
7. At least one measurable lesion (according to RECIST 1.1 criteria); Magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement accurately measured the diameter of ≥10mm, conventional CT scan to determine the diameter of at least 20mm.
8. No serious organic diseases of heart, lung, brain and other organs;
9. The functions of major organs and bone marrow are basically normal:

   1. Blood routine: white blood cells ≥ 4.0 x 109/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 80 x 109/L, hemoglobin ≥ 90g/L;
   2. International Standardized ratio (INR) and activated partial thrombin time (APTT) ≤1.5× upper limit of normal value (ULN);
   3. Liver function: serum total bilirubin ≤ 1.5 x ULN, ALT/AST ≤ 3 x ULN, serum total biliary red ≤ 1.5 x ULN after internal/external drainage for obstructive jaundice;
   4. Renal function: serum creatinine ≤ 1.5 x ULN, creatinine clearance (CCr) ≥ 50mL/min;
   5. Normal cardiac function, left ventricular ejection fraction (LVEF)≥50% by two-dimensional echocardiography;
10. Fertile male or female patients volunteered to use effective contraceptive methods, such as double screen contraceptives, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of the last study medication. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause or sterilization.

Those who met each of the above criteria were included in the study.

Exclusion Criteria:

The study proposal shall be excluded if any of the following criteria are met:

1. Participated in clinical trials of other antitumor drugs within 4 weeks before enrollment;
2. Prior treatment with VEGFR inhibitors or prior treatment with immune checkpoint inhibitors;
3. Patients with BRCA1/2 germ line mutation;
4. Patients with obstructive jaundice but failing to reach the expected yellow reduction;
5. Have had other malignancies within the past 5 years, other than basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
6. Patients who have had or currently have any brain metastases;
7. The investigators determined that liver metastases accounted for 70% or more of the total liver volume;
8. Had received any surgery (except biopsy) or invasive treatment or operation within 4 weeks prior to inclusion, and the surgical incision was not completely healed (except intravenous catheterization, puncture drainage, internal/external drainage for obstructive jaundice, etc.);
9. Uncontrolled pleural effusion, pericardial effusion or ascites requiring drainage;
10. Local antitumor therapy, such as hepatic artery interventional embolization, liver metastasis cryoablation or radiofrequency ablation, was received within 4 weeks before enrollment;
11. Electrolyte abnormalities identified by the investigator as clinically significant;
12. The patient has medically uncontrolled hypertension, as follows: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
13. Urine routine indicated urinary protein ≥2+ and 24-hour urinary protein volume > 1.0g;
14. Patients whose tumors are judged to be at high risk of invading vital blood vessels and causing fatal haemorrhage during the follow-up study;
15. Patients with significant evidence or history of bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, black feces, blood in stool), hemoptysis (within 4 weeks > 5 mL fresh blood); A history of hereditary or acquired bleeding or a coagulation disorder. Have clinically significant bleeding symptoms or definite bleeding tendency within 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.;
16. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; Electrocardiogram (ECG) showed a QT c interval ≥480 ms;
17. Active or uncontrolled severe infection (≥CTCAE grade 2 infection);
18. Unmitigated toxic reactions higher than CTCAE grade 2 or above due to any previous anticancer therapy, excluding grade 2 or less neurotoxicity due to alopecia, lymphocytopenia, and oxaliplatin;
19. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
20. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, the patient has a medical condition or condition that is reasonably suspected to be unsuitable for the use of the study drug (such as the presence of epileptic seizures requiring treatment), or which would interfere with the interpretation of the study results, or place the patient at high risk;
21. Known human immunodeficiency virus (HIV) infection; A known history of clinically significant liver disease, including viral hepatitis [active HBV infection must be ruled out as a known carrier of hepatitis B virus (HBV), i.e. positive HBV DNA (>1×104 copies/mL or >2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis;
22. The presence of any active, known or suspected autoimmune disease (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitaritis, hyperthyroidism, etc.);
23. Allergy or suspected allergy to the study drug or similar drug;
24. In the investigator's judgment, the patient had other factors that might affect the study results or lead to the termination of the study, such as alcoholism, drug abuse, other serious medical conditions (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, and family or social factors that would affect the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Defined as the time from the date of enrollment to the first documentation of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | The proportion of patients whose tumors have decreased by a certain degree and remained so for a specified duration, including cases of complete response (CR) and partial response (PR). Tumor objective response is assessed using RECIST v1.1
Overall survival | Overall survival (OS) refers to the duration from the date of enrollment to the date of death due to any cause.
Disease control rate | Defined as the proportion of evaluable patients with complete response (CR), partial response (PR), or stable disease (SD) as confirmed cases. At baseline, subjects must have measurable tumor lesions; responses are evaluated according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jin Xu, Principal Investigator — 180 1731 7267
Locations (1):
- Fudan University ShangHai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No